CLINICAL TRIAL: NCT04727528
Title: A Double-blind Randomized Placebo-controlled Parallel Design Multicenter Phase IIIb Study of the Effect of Sodium Zirconium Cyclosilicate (SZC) on Serum Potassium and Serum Bicarbonate in Patients With Hyperkalemia and Metabolic Acidosis Associated With Chronic Kidney Disease (NEUTRALIZE)
Brief Title: Study of the Effect of SZC on Serum Potassium and Serum Bicarbonate in Patients With Hyperkalemia and Metabolic Acidosis Associated With Chronic Kidney Disease
Acronym: NEUTRALIZE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to a higher than expected screen fail rate (83%) which lead to very low patient enrollment into the study. It should be noted that the decision to terminate the study is not related to safety concerns.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D9480C00022
Record Dates: First submitted 2020-12-22; First posted 2021-01-27 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Hyperkalaemia; Metabolic Acidosis; Chronic Kidney Disease
MeSH Terms: conditions — Hyperkalemia; Acidosis; Renal Insufficiency, Chronic | interventions — sodium zirconium cyclosilicate

STUDY DESIGN:
Intervention Model Description: NEUTRALIZE is a prospective, randomized, double-blind, placebo-controlled, parallel, multicenter, Phase IIIb study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Open-label correction phase (up to 48 hours) (Experimental): All eligible patients will receive SZC 10 g TID for up to 48 hours. Patients with POCT (Point-of-Care-Test) K+ ≥5.1 mmol/L after 24 hours will continue on SZC 10 g TID for another 24 hours. Patients who achieve normokalemia (defined as POCT K+ between 3.5 and 5.0 mmol/L inclusive) after receiving SZC 10 g TID for up to 48 hours will proceed to randomization.
  Patients with POCT K+ <3.5mmol/L at any time during the open-label phase will be withdrawn from study treatment and will be followed per protocol.
  Interventions: Drug: Sodium zirconium cyclosilicate; Drug: Placebo
- Randomized, placebo controlled phase (Day 2 or 3 to Day 29) (Experimental): Patients will be randomized to SZC 10 g QD or placebo 10 g QD. The dose of SZC/placebo will be titrated by increasing or decreasing the dose by 5 g increments at 1-week intervals to between 5 g every other day (QOD) and 15 g QD of the randomized phase to maintain normokalemia by POCT K+.
  Interventions: Drug: Sodium zirconium cyclosilicate; Drug: Placebo

INTERVENTIONS:
Drug: Sodium zirconium cyclosilicate — Investigational medicinal product
  Other Names: SZC
Drug: Placebo — Plabeco comparator

SUMMARY:
The main objective of this study is to evaluate the efficacy of SZC as compared to placebo in maintaining normal sK+ in patients with hyperkalemia and metabolic acidosis associated with CKD

DETAILED DESCRIPTION:
NEUTRALIZE is a prospective, randomized, double-blind, placebo-controlled, parallel, multicenter, Phase IIIb study to investigate the safety and efficacy of SZC in patients with hyperkalemia and low bicarbonate (metabolic acidosis ).

The study will be conducted in the United States (US) at approximately 35 investigative sites.

After screening on Day 1, all eligible patients will receive open-label SZC for up to 48 hours. Patients who achieve normokalemia within 48 hours will be randomized 1:1 into the double-blind randomized treatment phase to receive SZC or placebo. Study treatment will end with the Day 29 visit, which will be followed by a follow-up visit 7 days after the last administration of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years
* Participants who have CKD stage 3-5, not on dialysis.
* POCT K+ level >5 mmol/L to ≤5.9 mmol/L and POCT bicarbonate levels between 16-20 mmol/L inclusive prior to the first SZC dose on study Day 1
* Ability to have repeated blood draws or effective venous catheterization.
* Male and/or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent

Exclusion Criteria:

* Participants with pseudohyperkalemia.
* Dialysis requirement or anticipated by the investigator to require dialysis therapy within 1 month, history of renal transplant, or life expectancy less than 3 months.
* Cardiac arrhythmias requiring immediate treatment.
* Active or suspected diabetic ketoacidosis.
* POCT bicarbonate low enough to need emergency intervention or treatment as judged by the investigator.
* Acute/chronic worsening renal function (eg, ≥30% decline in eGFR) in the 3 months before screening.
* Current acute decompensated HF, hospitalization due to decompensated HF within 4 weeks prior to screening, or myocardial infarction (MI), unstable angina, stroke or transient ischemic attack (TIA) within 12 weeks prior to screening.
* Coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) or valvular repair/replacement within 12 weeks prior to screening or planned to undergo any of these operations.
* Symptomatic hypotension.
* Current exacerbation of chronic obstructive pulmonary disease (COPD)/asthma or hospitalization due to exacerbation of COPD/asthma within 4 weeks of screening.
* Severe constipation, bowel obstruction or impaction, including abnormal post-operative bowel motility disorders
* Active malignancy requiring treatment.
* History of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Patients with atrial fibrillation controlled by medication are permitted.
* QTcF (QT interval corrected by the Fridericia method) >550 msec.
* Active treatment (within 7 days prior to screening) with SZC, sodium bicarbonate, sodium polystyrene sulfonate, lactulose, or patiromer

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (28):
  - Research Site, Florence, Alabama
  - Research Site, Chula Vista, California
  - Research Site, Downey, California
  - Research Site, El Centro, California
  - Research Site, South Gate, California
  - Research Site, Victorville, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Coral Gables, Florida
  - Research Site, Columbus, Georgia
  - Research Site, Hinsdale, Illinois
  - Research Site, Kansas City, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Providence, Rhode Island
  - Research Site, Spartanburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, San Juan, Puerto Rico

REFERENCES:
- [Derived] Ash SR, Batlle D, Kendrick J, Oluwatosin Y, Kooienga L, Eudicone JM, Sundin AK, Guerrieri E, Fried LF. Sodium Zirconium Cyclosilicate in CKD, Hyperkalemia, and Metabolic Acidosis: NEUTRALIZE Randomized Study. Kidney360. 2024 Jun 1;5(6):812-820. doi: 10.34067/KID.0000000000000446. Epub 2024 Apr 16. PMID 38622759
- See also: CSRsynopsis_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00022&attachmentIdentifier=a2929651-81e2-4562-9b19-d5b5c9e0e34b&fileName=d9480c00022-study-synopsis-redacted.pdf&versionIdentifier=
- See also: SAP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00022&attachmentIdentifier=769d2427-ddee-4264-9488-9bf5c33d54f2&fileName=d9480c00022-sap-redacted-pdfa.pdf&versionIdentifier=
- See also: CSP_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480C00022&attachmentIdentifier=43a4bfc3-b957-4e04-a68b-3193a2d70a0b&fileName=d9480c00022-protocol-redacted-pdfa.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participants was randomized to the double-blind treatment phase in error but did not receive treatment. This participant is noted as not completing the open-label phase in the table below.
Groups:
- Sodium Zirconium Cyclosilicate (SZC): Open label phase: Three times daily (TID) 10 g SZC for up to 48 hours. Participants not achieving normokalemia or normokalemic at Day 2 continued in the open-label correction phase at 10 g SZC TID for an additional 24 hours and repeat point of care test on the next day (Day 3).
  Double-blind treatment phase: Double-blind TID 10 g SZC for up to 48 hours (not applicable in the open-label phase)
- Placebo: Open label phase: Three times daily (TID) 10 g SZC for up to 48 hours. Participants not achieving normokalemia or normokalemic at Day 2 continued in the open-label correction phase at 10 g SZC TID for an additional 24 hours and repeat point of care test on the next day (Day 3).
  Double-blind treatment phase: Double-blind placebo for up to 48 hours (not applicable in the open-label phase)
Period: Open-label Period
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Started (Participants entered open-label period and received treatment) | 39 (After screening on Day 1, all participants received open-label SZC for up to 48 hours, and then were randomized to double-blind treatment of SZC or placebo for 4 weeks.) | 0
Completed | 37 | 0
Not Completed | 2 | 0
Not completed — Did not meet randomization criteria for double-blind treatment phase | 1 | 0
Not completed — Randomized who did not receive treatment | 1 | 0
Period: Double-blind Treatment Phase
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Started | 17 (After the open-label period, participants were randomized into either the SZC or placebo group.) | 20 (After the open-label period, participants were randomized into either the SZC or placebo group.)
Completed | 16 | 15
Not Completed | 1 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Not completed — Missed doses whilst in hospital | 0 | 1
Not completed — Investigator decision to start rescue therapy for hyperkalemia | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Sodium Zirconium Cyclosilicate (SZC): Open label phase: Three times daily (TID) 10 g SZC for up to 48 hours. Participants not achieving normokalemia or normokalemic at Day 2 continued in the open-label correction phase at 10 g SZC TID for an additional 24 hours and repeat point of care test on the next day (Day 3).
  Double-blind treatment phase: Double-blind TID 10 g SZC for up to 48 hours
- Placebo: Open label phase: Three times daily (TID) 10 g SZC for up to 48 hours. Participants not achieving normokalemia or normokalemic at Day 2 continued in the open-label correction phase at 10 g SZC TID for an additional 24 hours and repeat point of care test on the next day (Day 3).
  Double-blind treatment phase: Double-blind placebo for up to 48 hours
- Total: Total of all reporting groups
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo | Total
Number analyzed (Participants) | 17 | 20 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (16.77) | 65.9 (11.13) | 63.3 (14.09)
Age, Customized [Number; unit: Participants] — Age at Screening Population: Full Analysis Set
  Participants
    >=85 | 0 | 0 | 0
    18-64 | 9 | 9 | 18
    65-84 | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Full Analysis Set
  Participants
    Female | 4 | 8 | 12
    Male | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    Hispanic or Latino | 6 | 4 | 10
    Not Hispanic or Latino | 11 | 16 | 27
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Full Analysis Set
  Participants
    American Indian or Alaskan Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Black or African American | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Other | 0 | 1 | 1
    White | 14 | 18 | 32
Diabetes status [Count of Participants; unit: Participants]
  No | 6 | 5 | 11
  Yes | 11 | 15 | 26
Chronic Kidney Disease (CKD) Status [Count of Participants; unit: Participants] — Stage 3a (G3a) - an eGFR of 45 to 59ml/min; Stage 3b (G3b) - an eGFR of 30 to 44ml/min; Stage 4 (G4) - an eGFR of 15 to 29ml/min; Stage 5 (G5) - an eGFR below 15ml/min, meaning the kidneys have lost almost all of their function
  Participants
    Stage 3 | 1 | 3 | 4
    Stage 4 | 14 | 8 | 22
    Stage 5 | 1 | 6 | 7
    Missing | 1 | 3 | 4
Chronic Heart Failure Status [Count of Participants; unit: Participants]
  No | 17 | 20 | 37
  Yes | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence (Yes/no) of Participants Having Normal Serum Potassium (sK+) Between 3.5 and 5.0 mmol/L Inclusive at End of Treatment (EOT) Without Need for Rescue Treatment for Hyperkalemia at Any Point During the Randomized Phase
Description: Response was defined as a subject having serum potassium (sK+) within 3.5-5.0 mmol/L at the EOT visit, and no use of rescue therapy for hyperkalaemia at any point during the randomized placebo-controlled period.
  Participants who used rescue therapy for hyperkalaemia at any point during the randomized placebo-controlled period were assigned a non-response. Participants who died prior to the EOT visit were treated as non-response. Participants who were lost to follow-up prior to the EOT visit had response treated as missing.
Time Frame: Day 1 of randomization phase to Day 29
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 1 | 15
  Response | 15 | 4
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Test type: Superiority; p = 0.001, Wald Chi-Squared test; Odds Ratio (OR) = 56.2, 95% CI 2-sided [5.6 to 563.6] — Logistic regression model included response status (response / non-response) as the dependent variable and randomized treatment as an independent factor

2. Secondary Outcome: Mean Serum Bicarbonate at Day 29
Description: Least-squares mean calculated with a repeated measures analysis of covariance model where the dependent variable was post randomization serum bicarbonate and with fixed terms for randomized treatment group and serum bicarbonate.
Time Frame: Day 29
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 16 | 17
mmol/L | 18.17 (0.58) | 16.52 (0.56)
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Difference between groups; Test type: Superiority; p = 0.050, t-test, 2 sided; Least-squares mean = 1.64, 95% CI 2-sided [-0.00 to 3.29], Standard Error of Mean 0.81

3. Secondary Outcome: Occurrence (Yes/no) of Participants Having an Increase in Serum Bicarbonate of Greater Than or Equal to 3 mmol/L From Baseline to EOT Without Need for Rescue Treatment for Metabolic Acidosis (Low Bicarbonate)
Description: Occurrence (yes/no) of participants having an increase in serum bicarbonate of greater than or equal to 3 mmol/L from baseline (Day 1) to EOT (Day 29) without need for rescue treatment for metabolic acidosis (low bicarbonate).
  Response was defined as a participant with an increase in serum bicarbonate greater than or equal to 3 mmol/L at the EOT visit without the need for rescue therapy for low bicarbonate. Participants who used rescue therapy for low bicarbonate at any point during the randomized placebo-controlled period had their last observation prior to rescue therapy carried forward. Participants who were lost to follow-up prior to the EOT visit had response treated as missing. Logistic regression model included response status (response / non-response) as the dependent variable and randomized treatment as an independent factor.
  Participants who died prior to the EOT visit were assigned a non-response.
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 10 | 16
  Response | 6 | 3
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Comparison between groups; Test type: Superiority; p = 0.153, Wald Chi-Squared test; Odds Ratio (OR) = 3.2, 95% CI 2-sided [0.6 to 15.8]

4. Secondary Outcome: Occurrence (Yes/no) of Participants Having Serum Bicarbonate ≥22 mmol/L
Description: Response was defined as a participant with an increase in serum bicarbonate greater than or equal to 22 mmol/L at the EOT visit without the need for rescue therapy for low bicarbonate. Participants who had used rescue therapy for low bicarbonate at any point during the randomized placebo-controlled period had their last observation prior to rescue therapy carried forward. Participants who died prior to the EOT visit were assigned a non-response. Participants who were lost to follow-up prior to the EOT visit had response treated as missing. Logistic regression model included response status (response / non-response) as the dependent variable and randomized treatment as an independent factor.
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 14 | 19
  Response | 2 | 0
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Comparison between groups; Test type: Superiority; p = 0.940, Wald Chi-Squared test; Odds Ratio (OR) = 57008.6, 95% CI 2-sided [lower limit 0.0] (The upper limit of the 95% confidence interval = 13124060000000000000000000000)

5. Secondary Outcome: Occurrence (Yes/no) of Participants Having an Increase in Serum Bicarbonate of Greater Than or Equal to 2 mmol/L From Baseline (Day 1) to EOT Without Need for Rescue Treatment for Metabolic Acidosis (Low Bicarbonate)
Description: Response was defined as a participant with an increase in serum bicarbonate greater than or equal to 2 mmol/L at the EOT visit and no use of rescue therapy for low bicarbonate at any point during the randomized placebo-controlled period. Participants who used rescue therapy for low bicarbonate at any point during the randomized placebo-controlled period had their last observation prior to rescue therapy carried forward. Participants who were lost to follow-up prior to the EOT visit had response treated as missing. Logistic regression model included response status (response / non-response) as the dependent variable and randomized treatment as an independent factor.
  Participants who died prior to the EOT visit were assigned a non-response.
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 8 | 13
  Response | 8 | 6
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Comparison between groups; Test type: Superiority; p = 0.271, Wald Chi-Squared test; Odds Ratio (OR) = 2.2, 95% CI 2-sided [0.5 to 8.6]

6. Secondary Outcome: Participants Having Normal sK+ at EOT and an Increase in Serum Bicarbonate of ≥3 mmol/L From Baseline Without Need for Rescue Treatment for Metabolic Acidosis (Low Bicarbonate) or Hyperkalemia
Description: Participants with normal sK+ between 3.5 and 5.0 mmol/L inclusive at EOT and increase in serum bicarbonate greater than or equal to 3 mmol/L from Day 1 without rescue treatment for metabolic acidosis (low bicarbonate) or hyperkalemia.
  Response was a participant with sK+ within 3.5-5.0 mmol/L and increase in serum bicarbonate greater than or equal to 3 mmol/L at the EOT visit and no use of rescue therapy for hyperkalaemia or low bicarbonate at any point during the randomized placebo-controlled period. Participants who used rescue therapy for low bicarbonate or HK during the randomized placebo-controlled period had last observation prior to rescue therapy carried forward. Participants lost to follow-up prior to EOT visit had response as missing. Logistic regression model included response status (response/non-response) as dependent variable and randomized treatment as an independent factor.
  Participants who died prior to the EOT visit were assigned a non-response.
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 10 | 18
  Response | 6 | 1
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Comparison between groups; Test type: Superiority; p = 0.039, Wald Chi-Squared test; Odds Ratio (OR) = 10.8, 95% CI 2-sided [1.1 to 102.8]

7. Secondary Outcome: Occurrence (Yes/no) of Patients Having a Normal sK+ Between 3.5 and 5.0 mmol/L Inclusive and Bicarbonate ≥22 mmol/L at Day 29 Without Need for Rescue Treatment for Hyperkalemia or Metabolic Acidosis (Low Bicarbonate)
Description: Response was defined as a participant with sK+ within 3.5-5.0 mmol/L and serum bicarbonate greater than or equal to 22 mmol/L at the EOT visit without the need for rescue therapy for hyperkalaemia or low bicarbonate. Participants who used rescue therapy for hyperkalaemia or low bicarbonate at any point during the randomized placebo-controlled period were assigned a non-response. Participants who were lost to follow-up prior to the EOT visit had response treated as missing. Logistic regression model included response status (response / non-response) as the dependent variable and randomized treatment as an independent factor.
  Participants who died prior to the EOT visit were assigned a non-response.
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  No response | 14 | 19
  Response | 2 | 0
  Missing | 1 | 1
Statistical Analysis 1: Comparison: Sodium Zirconium Cyclosilicate (SZC) vs Placebo; Comparison between groups; Test type: Superiority; p = 0.940, Wald Chi-Squared test; Odds Ratio (OR) = 57008.6, 95% CI 2-sided [lower limit 0.0] (The upper limit of the 95% confidence interval = 13124060000000000000000000000)

8. Secondary Outcome: Occurrence (Yes/no) of Participants Needing Rescue Treatment for Low Sodium Bicarbonate
Description: Occurrence (yes/no) of participants needing rescue treatment for low sodium bicarbonate any time during the randomized phase
Time Frame: Day 1 to Day 29 of randomization phase
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Sodium Zirconium Cyclosilicate (SZC) | Placebo
Number analyzed (Participants) | 17 | 20
Participants
  Rescue treatment required | 0 | 0
  Rescue treatment not required | 17 | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected at screening, during the open-label correction phase (Days 1 and 2), throughout the treatment period of the the randomization phase (Days 2 or 3 to 29 or 30 [end of treatment] or discontinuation), and during the follow up phase (Day 36 to 39).
Description: Adverse events were collected from the start of the open-label correction phase throughout the treatment period and including the follow-up period.
Groups:
- Open-Label Phase: Three times daily (TID) 10 g SZC for up to 48 hours. Participants not achieving normokalemia or normokalemic at Day 2 continued in the open-label correction phase at 10 g SZC TID for an additional 24 hours and repeat point of care test on the next day (Day 3).
- Sodium Zirconium Cyclosilicate (SZC) Double-blind Treatment Phase: Double-blind treatment phase: Double-blind TID 10 g SZC for up to 48 hours
- Placebo Double-blind Treatment Phase: Double-blind treatment phase: Double-blind placebo for up to 48 hours
Arm/Group | Open-Label Phase | Sodium Zirconium Cyclosilicate (SZC) Double-blind Treatment Phase | Placebo Double-blind Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/17 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/17 | 2/20
Other Adverse Events (participants affected / at risk) | 1/38 | 4/17 | 9/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Phase (N=38) | Sodium Zirconium Cyclosilicate (SZC) Double-blind Treatment Phase (N=17) | Placebo Double-blind Treatment Phase (N=20)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Phase (N=38) | Sodium Zirconium Cyclosilicate (SZC) Double-blind Treatment Phase (N=17) | Placebo Double-blind Treatment Phase (N=20)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (4)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to a screening failure rate higher than expected which led to early termination of the study, only 39 (17.0%) patients entered the open-label phase. Due to the early termination of the study and small sample size, the study was underpowered for the secondary efficacy endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years of completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04727528/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/28/NCT04727528/SAP_001.pdf